CLINICAL TRIAL: NCT01080768
Title: A Double Blind, Randomized, Parallel Study to Assess the Effects of Aliskiren/Amlodipine and Amlodipine Monotherapy on Ankle Foot Volume (AFV) in Patients naïve to Trial Drugs With Mild to Moderate Hypertension
Brief Title: Assessment of Aliskiren/Amlodipine and Amlodipine on Ankle Foot Volume (AFV) in Patients With Hypertension
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Publication of data from a similar study made the current study redundant.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSPA100A2201; 2009-014359-63 (EudraCT Number)
Record Dates: First submitted 2010-03-03; First posted 2010-03-04 (Estimated); Results first posted 2011-12-26 (Estimated); Last update posted 2011-12-26 (Estimated); Status verified 2011-11

CONDITIONS: Hypertension; Ankle Edema
Keywords: Pedal edema; hypertension; aliskiren; amlodipine
MeSH Terms: conditions — Hypertension | interventions — aliskiren; Amlodipine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Aliskiren/amlodipine + Placebo to amlodipine (Experimental): During the first week of active treatment, patients were instructed to take one tablet of aliskiren/amlodipine 150/5 mg and one capsule of placebo to amlodipine daily. For the 2nd to 4th week of active treatment, the patients were up-titrated to take 2 tablets of aliskiren/amlodipine 150/5 mg/day and 1 capsule of placebo to amlodipine.
  The patients were instructed to administer daily dose between 8:00 and 10:00 am preferably at the same time of the day.
  Interventions: Drug: Aliskiren/amlodipine; Drug: Placebo to Amlodipine
- Amlodipine + Placebo to aliskiren/amlodipine (Active Comparator): During the first week of active treatment, patients were instructed to take one capsule of amlodipine 5 mg and one tablet of placebo to aliskiren/amlodipine 150/5 mg daily. For the 2nd to 4th week of active treatment, the patients were up-titrated to take 1 capsule of amlodipine 10 mg/day and 2 tablets of placebo to aliskiren/amlodipine 150/5 mg/day.
  The patients were instructed to administer daily dose between 8:00 and 10:00 am preferably at the same time of the day.
  Interventions: Drug: Amlodipine; Drug: Placebo to Aliskiren/amlodipine

INTERVENTIONS:
Drug: Aliskiren/amlodipine — Aliskiren/amlodipine 150/5 mg/day
  Other Names: SPA100
  Arms: Aliskiren/amlodipine + Placebo to amlodipine
Drug: Amlodipine — Amlodipine 5 mg/day.
  Arms: Amlodipine + Placebo to aliskiren/amlodipine
Drug: Placebo to Aliskiren/amlodipine — Placebo to Aliskiren/amlodipine 150/10 mg/day
  Arms: Amlodipine + Placebo to aliskiren/amlodipine
Drug: Placebo to Amlodipine — Placebo to Amlodipine 5 mg/day
  Arms: Aliskiren/amlodipine + Placebo to amlodipine

SUMMARY:
The purpose of the present study was to evaluate the addition of aliskiren, to amlodipine can attenuate ankle edema formation in hypertensive patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients (male or female) with hypertension aged between 18-75 yrs.
* Patients not treated with amlodipine or no amlodipine in previous 1 year.
* Post-menopausal females

Exclusion Criteria:

* Patients unable to switch from prior hypertensive medication.
* Severe hypertension.
* Pregnant or nursing females.
* Patients with Type 1 or Type 2 diabetes mellitus
* History of immunodeficiency diseases, including a positive Human immunodeficiency virus (HIV) (Enzyme-linked immunosorbent assay [ELISA] and Western blot) test result.
* A positive Hepatitis B surface antigen (HBsAg) or Hepatitis C test result.

Other protocol-defined inclusion/exclusion criteria are applied

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2010-02; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (9):
- Netherlands (9):
  - Novartis Investigative Site, Beek en Donk
  - Novartis Investigative Site, Bosch
  - Novartis Investigative Site, Hoogwoud
  - Novartis Investigative Site, Lichtenvoorde
  - Novartis Investigative Site, Lieshout
  - Novartis Investigative Site, Poortvliet
  - Novartis Investigative Site, The Hague
  - Novartis Investigative Site, Utrecht
  - Novartis Investigative Site, Wildervank

RESULTS

PARTICIPANT FLOW:
Groups:
- Amlodipine+ Placebo to Aliskiren/Amlodipine: During the first week of active treatment, patients were instructed to take one capsule of amlodipine 5 mg and one tablet of placebo to aliskiren/amlodipine 150/5 mg daily. For the 2nd to 4th week of active treatment, the patients were up-titrated to take 1 capsule of amlodipine 10 mg/day and 2 tablets of placebo to aliskiren/amlodipine 150/5 mg/day.
  The patients were instructed to administer daily dose between 8:00 and 10:00 am preferably at the same time of the day.
Period: Overall Study
Arm/Group | Aliskiren/Amlodipine + Placebo to Amlodipine | Amlodipine+ Placebo to Aliskiren/Amlodipine
Started | 14 | 17
Completed | 12 | 16
Not Completed | 2 | 1
Not completed — Protocol Deviation | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aliskiren/Amlodipine + Placebo to Amlodipine | Amlodipine+ Placebo to Aliskiren/Amlodipine | Total
Number analyzed (Participants) | 14 | 17 | 31
Age Continuous [Mean (Standard Deviation); unit: years] | 55.4 (6.21) | 58.0 (4.49) | 56.8 (5.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 9 | 13 | 22

OUTCOME MEASURES:

1. Primary Outcome: Change in the Ankle Foot Volume (AFV) as Measured by Displacement Method
Description: AFV (mL) was measured using the principle of water displacement using a commercially available foot volumeter. The amount of water displaced in milliliters (mL) equals the volume of the foot/ankle. The study was terminated due to the publication of the results of a near identical study by Fogari et al. Hence, for the current study, no analysis was performed.
Time Frame: Baseline, 4 weeks
Population: The study was terminated due to the publication of the results of a near identical study by Fogari et al. Hence, for the current study, no analysis was performed.
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Aliskiren/Amlodipine + Placebo to Amlodipine | Amlodipine+ Placebo to Aliskiren/Amlodipine
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Groups:
- Aliskiren/Amlodipine and Placebo to Amlodipine: During the first week of active treatment, patients were instructed to take one tablet of aliskiren/amlodipine 150/5 mg and one capsule of placebo to amlodipine daily. For the 2nd to 4th week of active treatment, the patient up-titrated to take 2 tablets of aliskiren/amlodipine 150/5 mg/day and 1 capsule of placebo to amlodipine.
  The patients were instructed to administer daily dose between 8:00 and 10:00 am preferably at the same time of the day.
- Amlodipine and Placebo to Aliskiren/Amlodipine: During the first week of active treatment, patients were instructed to take one capsule of amlodipine 5 mg and one tablet of placebo to aliskiren/amlodipine 150/5 mg daily. For the 2nd to 4th week of active treatment, the patient up-titrated to take 1 capsule of amlodipine 10 mg/day and 2 tablets of placebo to aliskiren/amlodipine 150/5 mg/day.
  The patients were instructed to administer daily dose between 8:00 and 10:00 am preferably at the same time of the day.
Arm/Group | Aliskiren/Amlodipine and Placebo to Amlodipine | Amlodipine and Placebo to Aliskiren/Amlodipine
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/17
Other Adverse Events (participants affected / at risk) | 2/14 | 2/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aliskiren/Amlodipine and Placebo to Amlodipine (N=14) | Amlodipine and Placebo to Aliskiren/Amlodipine (N=17)
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Chest discomfort (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Otitis externa (Infections and infestations) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Dizziness (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.